CLINICAL TRIAL: NCT03562208
Title: Autologous Bone Marrow Transplant in Chronic Insulin Dependent Diabetic Patients Phase II Clinical Trial. Version: 1.3 - January 13, 2016
Brief Title: Autologous Bone Marrow Transplant in Chronic Insulin Dependent Diabetic Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Global Cell Med (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 132016
Record Dates: First submitted 2018-04-16; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus Progression; Diabetes Complications
Keywords: Diabetes Mellitus; Bone Marrow; Transplant
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Group 1 (50 patients): Patients treated with total bone marrow, in the protocol as a group treatment will analyze type OPEN: The patient knows the treatment, as the investigator and sponsor. All patients continue to receive the standard treatment with insulin and other medicines prescribed by your doctor.
  Group 2 (50 patients): Patient no treated, as a control group. All patients continue to receive the standard treatment with insulin and other medicines prescribed by your doctor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Adult Bone Marrow Stem Cells — Autologous Bone Marrow Stem Cells Transplant

SUMMARY:
Diabetes, recently declared a pandemic by the World Health Organization, is a risk factor for increased mortality and morbidity. Its multi-functional complications, in the short and long term, are a serious problems for the global public health. Millions of patients, the world over, suffer Diabetes, a chronic and degenerative disease without treatments today. America, and particularly the Caribbean and Central America Region, is seriously affected despite the efforts of the Public Health Systems. Caribbean Region presented nearly twice the incidence and prevalence of type 1 and type 2 diabetes when compared with the rest of the Americas. Today stem cells are emerging as a valid alternative of treatment. In vitro experiments with adult stem cells demonstrated their ability to migrate and differentiate into cells of different lineages. The bone marrow stem cells are safe, effective and have a lot of scientific evidence that supports the carrying out of clinical research in phases II and III. Our protocol is an Autologous Bone Marrow Stem Cell Transplantation, without immune suppression or cell cultures. Our hypothesis is that the stem cells will act as immune modulators, angiogenic and in a regenerative way stimulating quiescent stem cells and improving the metabolic control by endogenous secretion of insulin.

DETAILED DESCRIPTION:
Our clinical trial, authorized and controlled by the Government of Bahamas, offer safety data and effectiveness that encourage continued research. We will divide the patients into a treatment group and into a control group. We will control insulin daly dose, c peptide, A1C glycated hemoglobin and specific antibodies. Follow up two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic insulin dependent type 1 or 2 diabetes, with negative specific antibodies (Islets, GAD, E2) and low basal c peptide (Using C-peptide measurement (NV 0.9 mg / dl). Men and women, between 16 and 70 years old, derived voluntarily by their family doctors.

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
C Peptide | two years
  C Peptide measurement

SECONDARY OUTCOMES:
Insulin Daly Dose | Two years
A1C | Two Years

CONTACTS AND LOCATIONS:
Overall Officials: Desire Cox, MD, Study Director — National Stem Cell and Ethic Committee
Locations (1):
- Doctors Hospital, Nassau, New Providence District, The Bahamas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.stemcellbahamas.com